CLINICAL TRIAL: NCT02038621
Title: Phase II Clinical Study of the Maintenance Therapy of Capecitabine Afer the XELOX in Treatment of Advanced Gastric Cancer
Brief Title: The Maintenance Therapy of Capecitabine of Advanced Gastric Cancer
Acronym: GZH-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second People's Hospital of Sichuan (Other)
Responsible Party: Principal Investigator, Chengya Chou, Oncology physician, The Second People's Hospital of Sichuan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2ndSichuan; GZH-001
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Paclitaxel; Oxaliplatin; Capecitabine

ARMS (2):
- A (Experimental): Capecitabine: 1000mg/m^2 bid, days 1-14, every 3 weeks until progression/intolerance.
  Interventions: Drug: Paclitaxel; Drug: Oxaliplatin and Capecitabine
- B (Placebo Comparator): Observation until progression
  Interventions: Drug: Paclitaxel; Drug: Oxaliplatin and Capecitabine

INTERVENTIONS:
Drug: Paclitaxel
Drug: Oxaliplatin and Capecitabine — Before randomization,all enrolled patients underwent 3 cycles XELOX chemotheray. After patients' disease achieved CR\PR\SD,then randomized into this clinical trial.

SUMMARY:
To confirm the efficacy and safety of XELOX with capecitabine maintenance in treatment of advanced gastric cancer (AGC)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* male or female
* Patients with stage IV gastric cancer by pathology or cytology and imaging diagnosis , or after previous surgery or radiotherapy or chemotherapy in patients with stage IV gastric cancer progression , there RECIST criteria evaluable lesions ;
* ECOG performance status score 0-2 ;
* Expected survival time more than three months ;
* Adequate hematologic parameters and liver and kidney function ;
* Bone marrow : absolute neutrophil count (ANC) ≥ 1.5 × 109 / L, platelets ≥ 75 × 109 / L, hemoglobin ≥ 80g / L;
* Liver: bilirubin ≤ 1.5 times the upper limit of normal , ALT AST values ≤ 2.5 times the upper limit of normal ;
* Renal : serum creatinine ≤ ULN ;
* Informed consent of patients or their agents , and signed informed consent.

Exclusion Criteria:

* For patients allergic to capecitabine ;
* Patients with CNS metastases
* Undermine the integrity of the upper gastrointestinal tract , malabsorption syndrome , or unable to take oral medication ;
* Patients with coronary heart disease , angina , myocardial infarction , arrhythmia, cerebral thrombosis, stroke and other serious cardiovascular and cerebrovascular disease ;
* Or in combination with other anti-tumor therapy in patients participating in clinical trials of other interventions ;
* Pregnancy or breast-feeding patients , or fertility without taking adequate contraceptive measures were ;
* The researchers believe that this test is not suitable for those who participate .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
overall survival (OS) | from the date of randomization until death from any cause or up to 1 year
adverse events (AE) | from date of randomization to 28 days after the last chemo dosage
health-related quality of life (HRQOL | evaluate every 6 weeks from the date of randomization until 28 days after the last chemo dosage